CLINICAL TRIAL: NCT04362761
Title: A Phase 3b Open-label Extension Study Evaluating the Safety of Elexacaftor/Tezacaftor/Ivacaftor Combination Therapy in Cystic Fibrosis Subjects
Brief Title: A Study Evaluating the Long-Term Safety of Elexacaftor Combination Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX19-445-115; 2019-003455-11 (EudraCT Number)
Record Dates: First submitted 2020-04-22; First posted 2020-04-27 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX/TEZ/IVA (Experimental): Part A: Participants received elexacaftor (ELX) 200 milligram (mg) once daily (qd)/tezacaftor (TEZ)100 mg qd/ivacaftor (IVA)150 mg every 12 hours (q12h) in the treatment period for 48 weeks.
  Part B: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period up to 86 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination (FDC) tablet for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study evaluate the long-term safety and tolerability of elexacaftor (ELX)/tezacaftor (TEZ)/ ivacaftor (IVA) triple combination (TC) in participants with cystic fibrosis (CF) who are homozygous for F508del.

ELIGIBILITY:
Key Inclusion Criteria:

* Completed study drug treatment in parent study (VX18-445-109); or had study drug interruption(s) in parent study but completed study visits up to the last scheduled visit of the Treatment Period in the parent study

Key Exclusion Criteria:

* History of study drug intolerance in parent study

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- Australia (5):
  - The Prince Charles Hospital, Chermside
  - Institute for Respiratory Health, Nedlands
  - Telethon Kids Institute, Perth Children's Hospital, Nedlands
  - The Royal Children's Hospital, Parkville, VIC
  - Queensland Children's Hospital, South Brisbane
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Germany (6):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitaetsklinkum Koeln, CF-Studienzentrum, Cologne
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Universitatsklinikum Essen (AoR), Kinderklinik III, Abt. fur Pneumologie, Essen
  - Mukeviszidose-Zentrum am Universitatsklinikum Jena, Klinik fuer Kinder- und Jugendmedizin, Jena
  - Klinikum Innenstadt, University of Munich, München
- United Kingdom (16):
  - Belfast City Hospital, Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol Royal Hospital, Bristol
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter NHS Foundation Trust, Royal Devon and Exeter Hospital, Exeter
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - Leeds General Infirmary, Leeds
  - St. James University Hospital, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Sick Children, London
  - London and St Bartholomew's Hospital, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, The Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Queens Medical Center, Nottingham
  - All Wales Adult Cystic Fibrosis Centre, University Hospital Llandough, Penarth
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent research/clinical-trial-data-sharing.

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 2 parts, Part A and Part B. Participants from Part A also participated in Part B. The Participant flow was planned to be presented for the overall treatment arm.
Period: Part A (48 Weeks)
Arm/Group | ELX/TEZ/IVA
Started | 172
Completed | 159
Not Completed | 13
Not completed — Adverse Event | 2
Not completed — Withdrawal of consent (not due to AE) | 4
Not completed — Commercial drug is available for participant | 2
Not completed — Other | 5
Period: Part B (86 Weeks)
Arm/Group | ELX/TEZ/IVA
Started | 50 (Out of the 172 participants from Part A, only 50 participants participated in Part B of the study.)
Completed | 0
Not Completed | 50
Not completed — Commercial drug is available for participant | 46
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: Baseline data is based on the parent study baseline, which is defined as the most recent non-missing measurements collected before the first dose of the study drug in the treatment period of parent studies. Baseline data is presented for participants who received at least 1 dose of study drug in this study.
Groups:
- ELX/TEZ/IVA: Part A: Participants received ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 48 weeks.
  Part B: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period up to 86 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 172
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Baseline data were planned to be presented separately for Part A and Part B. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  years
    Part A | 27.9 (11.4)
    Part B: number analyzed (Participants) | 50
    Part B | 25.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and Part B. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  Participants
    Part A: Female | 87
    Part A: Male | 85
    Part B: number analyzed (Participants) | 50
    Part B: Female | 26
    Part B: Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and Part B. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  Participants
    Part A: Hispanic or Latino | 3
    Part A: Not Hispanic or Latino | 167
    Part A: Not collected per local regulations | 2
    Part B: number analyzed (Participants) | 50
    Part B: Hispanic or Latino | 1
    Part B: Not Hispanic or Latino | 49
    Part B: Not collected per local regulations | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and Part B. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  Participants
    Part A: White | 169
    Part A: Black or African American | 0
    Part A: Asian | 2
    Part A: American Indian or Alaska Native | 0
    Part A: Native Hawaiian or Other Pacific Islander | 0
    Part A: White, Asian | 1
    Part A: Not collected per local regulations | 0
    Part B: number analyzed (Participants) | 50
    Part B: White | 50
    Part B: Black or African American | 0
    Part B: Asian | 0
    Part B: American Indian or Alaska Native | 0
    Part B: Native Hawaiian or Other Pacific Islander | 0
    Part B: White, Asian | 0
    Part B: Not collected per local regulations | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Safety and Tolerability as Assessed by Number of Participants With Treatment- Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to Week 52
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: ELX/TEZ/IVA: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 48 weeks.
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 172
Participants
  Participants with TEAEs | 160
  Participants with SAEs | 26

2. Primary Outcome: Part B: Safety and Tolerability as Assessed by Number of Participants With Treatment- Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to Week 86
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: ELX/TEZ/IVA: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg qd in the treatment period up to 86 weeks.
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 50
Participants
  Participants with TEAEs | 50
  Participants with SAEs | 8

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 52 for Part A, Day 1 up to Week 86 for Part B
Description: MedDRA 24.0 for Part A and MedDRA 25.1 for Part B.
Groups:
- Part A: ELX/TEZ/IVA: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg qd in the treatment period for 48 weeks.
Arm/Group | Part A: ELX/TEZ/IVA | Part B: ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/50
Serious Adverse Events (participants affected / at risk) | 26/172 | 8/50
Other Adverse Events (participants affected / at risk) | 127/172 | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=172) | Part B: ELX/TEZ/IVA (N=50)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Vascular device occlusion (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 8 | 5
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Forced expiratory volume decreased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Dissociative disorder (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=172) | Part B: ELX/TEZ/IVA (N=50)
Abdominal pain (Gastrointestinal disorders) | 16 | 3
Abdominal pain upper (Gastrointestinal disorders) | 12 | 2
Constipation (Gastrointestinal disorders) | 10 | 4
Diarrhoea (Gastrointestinal disorders) | 13 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 9 | 1
Vomiting (Gastrointestinal disorders) | 8 | 3
Fatigue (General disorders) | 13 | 1
Malaise (General disorders) | 3 | 3
Pyrexia (General disorders) | 7 | 8
Immunisation reaction (Immune system disorders) | 0 | 7
COVID-19 (Infections and infestations) | 2 | 17
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 17 | 21
Influenza (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 28 | 16
Upper respiratory tract infection (Infections and infestations) | 10 | 11
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3
Vaccination complication (Injury, poisoning and procedural complications) | 24 | 0
Alanine aminotransferase increased (Investigations) | 9 | 1
Aspartate aminotransferase increased (Investigations) | 11 | 0
Blood bilirubin increased (Investigations) | 11 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4
Dizziness (Nervous system disorders) | 11 | 0
Headache (Nervous system disorders) | 42 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 19 | 5
Rash (Skin and subcutaneous tissue disorders) | 12 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT04362761/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT04362761/SAP_001.pdf